CLINICAL TRIAL: NCT06880471
Title: Effects of TheraCal PT, Biodentin, and MTA on Postoperative Pain After Full Pulpotomy in Permanent Teeth With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Postoperative Pain After Full Pulpotomy With TheraCal PT, Biodentin, and MTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Fatos Albayrak, Assistant Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-03/06; DİŞ-2024-327 (Other Grant/Funding Number: Sivas Republic University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-01-21; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ProRoot MTA Application Procedure (Active Comparator): The coronal pulp tissue of the tooth will be removed using a high-speed sterile diamond bur. Then, hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl for 2 minutes, and this procedure may be repeated up to 3 times (totaling 6 minutes) if necessary. After confirming bleeding control, ProRoot MTA material will be placed at the canal openings. Following a waiting period of 15 minutes, Resin Modified Glass Ionomer Cement (RMCIS) will be applied as the base material (Vitrebond, 3M; ESPE) in a thin layer. Finally, restorative treatment of the tooth will be performed to complete the procedure.
  Interventions: Biological: TheraCal PT pulpotomy; Biological: Biodentine pulpotomy
- Biodentine Application Procedure (Active Comparator): After the coronal pulp tissue of the tooth is removed using a high-speed sterile diamond bur, hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl for 2 minutes, and this may be repeated up to 3 times (for a total of 6 minutes) if necessary. Once bleeding control is established, Biodentin material will be placed at the canal openings. After a waiting period of 12 minutes according to the manufacturer's instructions, Resin Modified Glass Ionomer Cement (RMCIS) will be applied as a base material (Vitrebond, 3M; ESPE) in a thin layer. Finally, restorative treatment of the tooth will be performed to complete the procedure.
  Interventions: Biological: TheraCal PT pulpotomy; Biological: MTA pulpotomy
- TheraCal PT Application Procedure (Active Comparator): After the coronal pulp tissue of the tooth is removed using a high-speed sterile diamond bur, hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl for 2 minutes, and this may be repeated up to 3 times (totaling 6 minutes) if necessary. Once bleeding control is established, TheraCal PT material will be placed. According to the manufacturer's instructions, after a 10-second irradiation period, Resin Modified Glass Ionomer Cement (RMCIS) will be applied as a base material (Vitrebond, 3M; ESPE) in a thin layer. Finally, restorative treatment of the tooth will be performed to complete the procedure.
  Interventions: Biological: MTA pulpotomy; Biological: Biodentine pulpotomy

INTERVENTIONS:
Biological: TheraCal PT pulpotomy — After the coronal pulp tissue is removed using a high-speed sterile diamond bur and bleeding control is achieved, TheraCal PT material will be placed. According to the manufacturer's instructions, the irradiation time is 10 seconds. It is dual-cure. Its content is based on calcium silicate modified with resin.
  Arms: Biodentine Application Procedure; ProRoot MTA Application Procedure
Biological: MTA pulpotomy — After the coronal pulp tissue is removed using a high-speed sterile diamond bur and bleeding control is achieved, ProRoot MTA material will be placed. After waiting for 15 minutes for it to set, the restorative treatment will be performed. MTA consists of the main components: tricalcium silicate, dicalcium silicate, tricalcium aluminate, tricalcium oxide, silicate oxide, and calcium sulfate dihydrate.
  Arms: Biodentine Application Procedure; TheraCal PT Application Procedure
Biological: Biodentine pulpotomy — After the coronal pulp tissue is removed using a high-speed sterile diamond bur and bleeding control is achieved, Biodentin material will be placed. After waiting for 12 minutes according to the manufacturer's instructions for it to set, the restorative treatment will be performed. Biodentin is a two-component material. The powder primarily consists of tricalcium silicate.
  Arms: ProRoot MTA Application Procedure; TheraCal PT Application Procedure

SUMMARY:
In this study, the researchers will evaluate the effect of three highly biocompatible materials-TheraCal PT (ThPT), Biodentin, and MTA-on postoperative pain in permanent teeth affected by deep caries and symptomatic irreversible pulpitis.

Participants:

The study will include 51 participants aged between 18 and 45 years who are systemically healthy.

Methodology:

Pulpotomy Procedure:

Pulpotomy will be performed on the lower first molar tooth of each participant. The teeth will be randomly divided into three groups, with 17 participants in each group. Coronal pulp tissue will be removed using a high-speed sterile diamond bur. Hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl, and this procedure may be repeated up to three times (totaling 6 minutes) if necessary.

Use of Biocompatible Materials:

After achieving hemostasis, one of the three biocompatible materials (TheraCal PT, Biodentin, or MTA) will be applied to the canal access. Participants will be prescribed NSAIDs.

Pain Assessment:

Preoperative Assessment : The pain intensity of participants will be recorded before treatment.

Postoperative Assessment : Participants will report their pain intensity at the 6th, 24th, 48th, and 72nd hours and on the 7th day using the Visual Analogue Scale (VAS). Participants will return with their VAS charts for evaluation at the end of one week.

Comparative Analysis:

The primary outcome will be a comparative evaluation of postoperative pain intensity values among the three different materials used in pulpotomy treatment. This study aims to provide valuable information on the effectiveness of various biocompatible materials in postoperative pain management and to contribute to improving clinical decision-making processes in endodontic treatments.

DETAILED DESCRIPTION:
The ethical approval for our study has been obtained from the Clinical Research Ethics Committee of Sivas Cumhuriyet University. The experimental phase of the study will be conducted at the Department of Endodontics, Faculty of Dentistry, Sivas Cumhuriyet University.

Patient Selection Criteria:

Participants aged between 18 and 45, who present with findings of irreversible pulpitis in the lower first molar tooth and apply to the Department of Endodontics, Faculty of Dentistry, Sivas Cumhuriyet University, will be included in the study.

In this study:

When α=0.05, β=0.10, and 1-β=0.90 were set, it was decided to include 17 teeth in each group, and the power of the test was found to be p=0.90948.

Statistical Method:

The data obtained from our study will be recorded in the SPSS 22.0 program. When the assumptions for parametric tests (Shapiro-Wilk) are met, one-way ANOVA will be used to compare measurements obtained from two or more independent groups. If differences are found, a Tukey test will be performed to determine which groups differ. If the parametric assumptions are not met, the Kruskal-Wallis test will be applied, and the Mann-Whitney U test will be used to identify the differing groups. The data will be presented in tables, including arithmetic mean, standard deviation, median, minimum-maximum values, and the error level will be set at 0.05.

Inclusion Criteria for the Study:

Age between 18 and 45 years, Absence of systemic disease, Apical periodontitis findings may be present or not, Symptoms of irreversible pulpitis must be present, The apex of the tooth must be closed, Pulp sensitivity tests (cold test and electric pulp test) must respond positively, Periodontal pocket depth and mobility must be within normal limits, Rubber dam isolation must be provided for the tooth to be treated, Restorative treatment of the tooth must be possible, The patient's mouth opening must be sufficient.

Exclusion Criteria from the Study:

Presence of any systemic disease (including conditions requiring prophylaxis), Presence of mental or psychiatric disorders, Presence of any allergic condition, Use of painkillers in the last 12 hours before the procedure or antibiotics in the last week, Loss of tooth structure that cannot be restoratively treated, Presence of a fistula tract or abscess, Negative response to pulp sensitivity tests (cold test and electric pulp test), No bleeding in the pulp or failure to achieve hemostasis within 6 minutes after total pulpotomy, Open apex, Advanced canal calcification observed on periapical radiography, Presence of internal or external root resorption.

After clinical and radiographic examinations, pulpal and periapical diagnosis will be established before the procedure. A diagnostic periapical radiograph will be taken using a film holder with the parallel technique to visualize the depth of the carious lesion and evaluate the periapical area. All patients will be informed about treatment details, materials used, possible complications, follow-up dates, and alternative treatment options. A written consent form will be obtained from patients indicating alternative options for root canal treatment, tooth extraction, or withdrawal from treatment. Prior to treatment, the pre-operative pain values of participants will be recorded. The pulpotomy procedure will be carried out according to the following protocol:

Anesthesia : Anesthesia will be provided using 4% articaine with 1:100,000 epinephrine. The tooth will be isolated with a rubber dam. The tooth designated for pulpotomy will be disinfected using 5% NaOCl before the procedure. After cleaning the caries, the exposed coronal pulp tissue will be amputated to the level of the canal orifices using a high-speed sterile diamond bur. Pulp vitality will be assessed visually by checking for bleeding at each canal orifice. Hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl for 2 minutes, and this will be repeated up to three times (for a total of 6 minutes) if necessary.

After achieving hemostasis, the pulp capping material will be randomly selected from ProRoot MTA (Denstply), Biodentin (Septodont), or TheraCal PT (ThPT, Bisco Inc) using www.randomizer.org. The application of materials will be performed according to the manufacturer's instructions.

Applications:

ProRoot MTA Application :

Coronal pulp tissue will be removed using a high-speed sterile diamond bur. Then, hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5 % NaOCl for 2 minutes, and this will be repeated up to three times (totaling 6 minutes) if necessary. After confirming bleeding control, the ProRoot MTA material will be placed at the canal openings. After a waiting period of 15 minutes, a thin layer of Resin Modified Glass Ionomer Cement (Vitrebond, 3M; ESPE) will be applied as the base material. Finally, the tooth will receive restorative treatment to complete the procedure.

Biodentin Application :

Coronal pulp tissue will be removed using a high-speed sterile diamond bur, and hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl for 2 minutes, repeated up to three times (totaling 6 minutes) if necessary. After confirming bleeding control, the Biodentin material will be placed at the canal orifices. According to the manufacturer's instructions, after a waiting period of 12 minutes, a thin layer of Resin Modified Glass Ionomer Cement (Vitrebond, 3M; ESPE) will be applied as the base material. Finally, the tooth will receive restorative treatment to complete the procedure.

TheraCal PT Application :

After the coronal pulp tissue is removed using a high-speed sterile diamond bur, hemostasis will be achieved by applying gentle pressure with a cotton pellet soaked in 2.5% NaOCl for 2 minutes, and this will be repeated up to three times (totaling 6 minutes) if necessary. After confirming bleeding control, the TheraCal PT material will be placed. Following a 10-second irradiation period according to the manufacturer's instructions, a thin layer of Resin Modified Glass Ionomer Cement (Vitrebond, 3M; ESPE) will be applied as the base material. Finally, the tooth will receive restorative treatment to complete the procedure.

Monitoring and Pain Assessment:

After the treatment, participants will be asked to fill out the Visual Analog Scale (VAS) chart to determine the severity of pain. Participants will be instructed to indicate their pain intensity at that moment on the VAS chart, marking between 0-100 mm, for the 6th hour, 24th hour, 48th hour, 72nd hour, and 7th day. Participants will be contacted in person or by phone for reminders over a 7-day period regarding when to fill out the form. At the end of the week, participants will be asked to return to the clinic with their VAS charts for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age range should be between 18 and 45,
2. Systemic disease should be absent,
3. Apical periodontitis findings may or may not be present,
4. Irreversible pulpitis symptoms should be present,
5. The apex of the tooth should be closed,
6. Pulp sensitivity tests (cold test and electric pulp test) should respond positively,
7. Periodontal pocket depth and mobility should be within normal limits,
8. Rubber dam isolation should be provided for the tooth to be treated,
9. Restorative treatment of the tooth should be performed,
10. The patient's mouth opening should be sufficient.

Exclusion Criteria:

1. The patient has any systemic disease (including conditions requiring prophylaxis),
2. The patient has mental or psychiatric disorders,
3. The patient has any allergic condition,
4. The patient has used painkillers in the last 12 hours before the procedure and antibiotics in the last week,
5. There is a loss of material in an amount that cannot be restoratively treated,
6. The presence of a fistula tract or abscess,
7. A negative response to pulp sensitivity tests (cold test and electric pulp test),
8. No bleeding in the pulp or failure to achieve hemostasis within 6 minutes after total pulpotomy,
9. The apex is open,
10. Advanced canal calcification is observed on periapical radiography,
11. The presence of internal or external root resorption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of postoperative pain caused by TheraCal PT, Biodentin and MTA application at 6, 24, 48, 72 hours and 7 days | 6, 24, 48, 72 hours and 7 days
  In the study, TheraCal PT, Biodentin, and MTA materials will be applied to teeth with irreversible pulpitis. Preoperative pain values and postoperative pain values at 6, 24, 48, 72 hours and on the 7th day will be recorded. The preoperative and postoperative values of TheraCal PT, Biodentin, and MTA materials will be evaluated comparatively.

OTHER OUTCOMES:
Primary Outcome Measure Secondary Outcome Measure Other Pre-Specified Outcome | The VAS questionnaire will assess postoperative pain at 6, 24, 48, 72 hours and 7 days.
  Postoperative pain will be assessed using the Visual Analog Scale (VAS) by the participants. Participants will mark the point on the line that they believe represents their current condition. The VAS score is determined by measuring the distance in millimeters from the left end of the line to the point marked by the participant using a ruler, resulting in a score between 0 and 100. Post-treatment pain intensity is classified as none (0-4 mm), mild (5-44 mm), moderate (45-74 mm), or severe (75-100 mm).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Dentistry, Sivas Cumhuriyet University, Sivas
  - Sivas Republic University Faculty of Dentistry, Sivas